CLINICAL TRIAL: NCT04845906
Title: A 7 Day Adhesive Device Wear Study to Evaluate BD StatLock™ Devices
Status: Completed | Type: Observational
Sponsor: Becton, Dickinson and Company (Industry)
Responsible Party: Sponsor
Other Study IDs: MDS-21STLOCK001
Record Dates: First submitted 2021-04-09; First posted 2021-04-15 (Actual); Last update posted 2021-09-08 (Actual); Status verified 2021-09

CONDITIONS: Peripheral Intravenous Catheter Stabilization

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Healthy volunteers: There will be 4 separate StatLock™ devices being tested, which will be randomly applied to the participants on their inner (ventral) forearms. Each participant will have 2 separate devices applied, one to each arm. Those participants who have the StatLock ™ Arterial Plus, StatLock™ Dialysis II, or the StatLock IV Select, will also have the foam strip applied.
  Interventions: Device: StatLock™ Catheter Stabilization Device and the StatLock™ stabilization device accessory (Foam Strip)

INTERVENTIONS:
Device: StatLock™ Catheter Stabilization Device and the StatLock™ stabilization device accessory (Foam Strip) — Each participant will have 2 separate devices applied, one to each arm, with or without a Foam Strip.The participant will also wear a dressing over top of a StatLock™ compatible catheter, which will be connected to an extension set. For this study, the catheter will not be inserted into the study participant but instead will be shortened or modified and placed on the skin and secured with the StatLock™ Stabilization Device. The use of the catheters, extension set, and the dressing represents how the device would be used in a clinical setting.
  Other Names: StatLock™ Pro- SLP001; StatLock™ IV Select- IV0521CE; StatLock™ Arterial Plus- ART0222CE; StatLock™ Dialysis II- VDS2; Foam Strip- SL0100 (StatLock™ Stabilization Device Accessory)

SUMMARY:
This study is a prospective healthy human volunteer wear study to evaluate the safety and performance of the StatLock™ Catheter Stabilization Device and the StatLock™ stabilization device Accessory (Foam Strip) and to meet the design input requirements.

DETAILED DESCRIPTION:
This is a healthy human wear study of a minimum of 100 study participants who will wear the StatLock™ Catheter Stabilization Device and the StatLock™ stabilization device accessory (Foam Strip). Participants will report to the research center, on Day 0 to have their skin assessed by the investigator, clinician, and/or designee. On Day 0 the participants will have the StatLock™ Catheter Stabilization Devices and the foam strip applied. There will be 4 separate StatLock™ devices being tested, which will be randomly applied to the participants on their inner (ventral) forearms. Each participant will have 2 separate devices applied, one to each arm. Those participants who have the StatLock ™ Arterial Plus, StatLock™ Dialysis II, or the StatLock IV Select , will also have the Foam Strip applied.

The participant will also wear a dressing over top of a StatLock™ compatible catheter, which will be connected to an extension set. For this study, the catheter will not be inserted into the study participant but instead will be shortened or modified and placed on the skin and secured with the StatLock™ Stabilization Device. The catheter tip will be marked with indelible ink, to assess for any catheter movement. The use of the catheters, extension set, and the dressing represents how the device would be used in a clinical setting.

Once the devices are applied the participant will have the skin assessed (using a modified Draize Scale) by the investigator, clinician, and/or designee on Day 0. The participant will wear the devices at home for 1 week and will return on Day 7 for a skin assessment, evaluation of pad and foam strip lift, and catheter movement, evaluation of pain, and removal of the devices by the investigator, clinician, and/or designee. On Day 8, there may be a phone call and/or video call with the participant to review the skin condition of the site where the device was removed from.

ELIGIBILITY:
Inclusion Criteria:

* Any healthy human, 14 years of age or older, regardless of gender (Note: Consent of guardian or parent may be required for patients who are under 18 years of age).
* If they provide written and informed consent.
* Expected to be available for observation from consent, to the application on Day 0, and then removal of the StatLock™ Catheter Stabilization Device on Day 7, and for a follow up phone and/or video call on Day 8 for a skin assessment.
* Participant agrees to maintain a diary from device application, Day 0, through device removal, Day 7.
* Agree to keep the StatLock™ Catheter Stabilization Device, ancillary products, and site dry throughout the study
* Agrees to not use moisturizers, lotions, or any product labeled moisturizing for the duration of the study, at or around the site where the devices will be applied (inner (ventral) forearm).

Exclusion Criteria:

* If their skin was burned or scarred at the insertion site, or has any other skin condition which may affect the adherence and/or interpretation of the study results.
* If they have a known allergy to the study products (known tape or adhesive allergy).
* Has a medical condition which may prevent him or her from completing the study or place the study participant at undue risk.

Min Age: 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Potential participants will be recruited from healthy volunteer participant pools identified and/or held by the study site(s).
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2021-07-13 (Actual); Primary Completion 2021-08-23 (Actual); Study Completion 2021-08-23 (Actual)

PRIMARY OUTCOMES:
Percent lift of the StatLock™ Catheter Stabilization Device Pad at Day 7 | Day 7
  Device pad lift will be assessed using a Visual Analog Scale, ranging from 0 - Fully adhered to 100 - Device absent. When the percent lift at day 7 is >50%, it is considered a failure.
Percent of Device Movement of the StatLock™ Catheter Stabilization Device at Day 7 | Day 7
  The percent of device movement of the catheter will be assessed using a Visual Analog Scale from 0 (no movement) to 100 (completely displaced).
Ease of Removal of the StatLock™ Catheter Stabilization Device | Day 7
  Ease of removal will be assessed using a 100 mm Visual Analog Scale where 0 is very easy to remove and 100 is very difficult to remove.
Percent of participants with erythema score ≥ 2 | Day 7
  Erythema score will be assessed using a modified Draize scale with scores ranging from 0 to 3, as follows: 0 - no visible reaction; 0.5 - Doubtful or negligible erythema reaction; 1.0 - mild or just perceptible macular erythema reaction in a speckled/follicular, patchy or confluent pattern (slight pinking); 2.0 - Moderate erythema reaction in a confluent pattern (definite redness); 3 - Strong or brisk erythema reaction that may spread beyond the test site).

SECONDARY OUTCOMES:
Percent lift of the Foam Strip (StatLock™ Stabilization Device Accessory) at Day 7 | Day 7
  The percent lift of the foam strip will be assessed using a Visual Analog Scale ranging from 0 (fully adhered) to 100 (device accessory absent).
Ease of Removal of the StatLock™ Stabilization Device Foam Strip | Day 7
  The ease of removal will be assessed using a 100 mm Visual Analog Scale where 0 is very easy to remove and 100 is very difficult to remove.
Level of pain upon removal of the StatLock™ Catheter Stabilization Device | Day 7
  Pain upon removal of the device will be assessed using a 100 mm Visual Analog Scale where 0 is no pain and 100 is unbearable pain.

OTHER OUTCOMES:
Rate of StatLock™ Catheter Stabilization device-related adverse events | Day 0 to Day 8
  Rate of device-related adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Casser, MD, Principal Investigator — TKL Research, Inc.; Gary Grove, PhD, Principal Investigator — Dermico, LLC
Locations (2):
- United States (2):
  - TKL Research, Inc, Fair Lawn, New Jersey
  - Dermico, LLC, Broomall, Pennsylvania